CLINICAL TRIAL: NCT00452270
Title: A Double-Blind, Randomized, Parallel Group, Placebo Controlled Study, Evaluating the Decongestant Effect, Time to Onset, Duration of Effect and Impact on Sleep and General Well-Being of Xylometazoline in Subjects With a Common Cold
Brief Title: Decongestant Effect, Timing of Effect and Impact on Sleep and General Well-Being of Xylometazoline in Subjects With a Common Cold
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OTCS-CE-301
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2007-05-03 (Estimated); Status verified 2007-05

CONDITIONS: Common Cold
Keywords: Common cold, xylometazoline
MeSH Terms: conditions — Common Cold | interventions — xylometazoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Xylometazoline

SUMMARY:
The aim of this study is to characterize the time profile of the decongestant properties of xylometazoline and to investigate its effect on sleep, general well-being and smell/taste.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Have had moderate common cold symptoms for less than 36 hours.

Exclusion Criteria:

* Congested/runny nose for more than two continuous weeks in the previous 12 months
* Deviated septum or nasal polyps
* Recent use of antibiotics
* Recent sinusitis

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2007-03; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the decongestant effect of xylometazoline in subjects with
common cold compared to placebo treatment by means of rhinomanometry over a period of 12 hours.

SECONDARY OUTCOMES:
To measure the peak subjective effect, time to onset of subjective relief of nasal obstruction
and duration of relief of nasal obstruction

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Investigative Site, Cardiff, Wales, UK, Principal Investigator
Locations (1):
- Novartis Investigative Site, Cardiff, Wales, United Kingdom